CLINICAL TRIAL: NCT07154381
Title: Monocentric Observational Trial for Florbetaben PET/MRI Hybrid Imaging in Patients With Cardiac Amyloidosis
Brief Title: Hybrid Florbetaben PET/MRI for Imaging of Cardiac Amyloidosis
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-8798-BO
Record Dates: First submitted 2025-05-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Amyloidosis
Keywords: PET/MRI; Florbetaben
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Amyloidosis: Oberservation of patients with proven cardiac amyloidosis and Florbetaben PET/MRI as part of diagnostic work up

SUMMARY:
Exploration of prognostic parameters in 18F-Florbetaben PET/MRI in patients with cardiac amyloidosis. The clinical endpoints are defined as occurence of major adverse cardiac events (MACE) in amyloidosis patients. Additionally, MACE outcome stratified by PET parameters will be evaluated and individual parameters of the imaging techniques will be compared to each other (PET, MRI or echocardiography).

DETAILED DESCRIPTION:
The aim of the study is to investigate the value of hybdrid imaging using 18F-Florbetaben PET/MRI for detecting prognostically relevant disease markers in patients with cardiac amyloidosis. The clinical endpoints are defined as occurence of major adverse cardiac events (e.g. hospitalizations due to heart failure, cardiovascular mortality, implantation of cardioverters etc.) in PET positive and negative patients.

Additionally, MACE outcome stratified by PET parameters will be evaluated and individual parameters of the imaging techniques will be compared to each other. CMR imaging will focused on LGE presence, ECV, native T1 mapping and echocardiography on commonly used markers includiging EF, Strain, E/e' and other functional parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* proven Amyloidosis (ATTR or AL)
* Women: negative pregnancy test less than weeks prior imaging.

Exclusion Criteria:

* Patients receiving amyloidosis-specific treatment prior study inclusion.
* Patients participating in other clinical trails for treatment of Amyloidosis.
* Pregnancy
* Contraindiactions for MRI (eGFR<30ml/min/1.73m2; gadolinium allergy; metallic implants or device not suited for 3T MRI).
* inability of consent
* Refusal of consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven amyloidosis with no competing amyloidosis treatments, willing and capable of undergoing Florbetaben PET/MRI.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Occurence of MACE | 36 Months
  Occurence of MACE, MACE defined as All-cause of Death or Hospitalization due to heart failure, implantation of a cardioverter defibrillator or other urgent cardiovascular intervention.

SECONDARY OUTCOMES:
MACE free survival by optimal tracer retention index for MACE | 36 Months
  MACE free survival by optimal tracer retention index (RI), threshold defined by ROC analysis for prediction of MACE.
MACE free survival by optimal SUV threshold for MACE | 36 Months
  MACE free survival by optimal standardized uptake value (SUV), threshold defined by ROC analysis for prediction of MACE.
MACE free survival by optimal retention index for AL-Amyloidosis | 36 Months
  MACE free survival by optimal SUV, threshold defined by ROC analysis for prediction of AL-Amyloidosis.
MACE free survival by optimal PET based threshold for AL-Amyloidosis | 36 Months
  MACE free survival by optimal tracer retention index (RI) defined by ROC analysis for prediction of AL-Amyloidosis.
Hazard Ratios for SUV | 36 Months
  Hazard Ratios for SUV PET parameters by univariate regression analysis
Hazard Ratios for retention index | 36 Months
  Hazard Ratios for tracer retention index by univariate regression analysis
Hazard Ratios for tracer washout | 36 Months
  Hazard Ratios for tracer washout by univariate regression analysis
Hazard Ratios for visual PET positivity | 36 Months
  Hazard Ratios for visual PET positivity defined by clear higher-than-background tracer uptake at 40-60 min post. injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear medicine, University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No